CLINICAL TRIAL: NCT03374787
Title: Single Center Evaluation of a Sound Processor for a Transcutaneous System
Brief Title: Evaluation of Sound Processor for a Transcutaneous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: C58
Record Dates: First submitted 2017-12-04; First posted 2017-12-15 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Conductive Hearing Loss; Mixed Hearing Loss
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fusion sound processor (Experimental): The sound processor picks up the sound and transfer it to the implant that convert the sound to vibrations that are transmitted to the inner ear.
  Interventions: Device: Fusion Sound Processor

INTERVENTIONS:
Device: Fusion Sound Processor — Sound Processor

SUMMARY:
A single center study evaluating the performance of an externally worn sound processor for a transcutaneous bone anchored hearing system using audiological outcomes measures such as aided thresholds and speech intelligibility and self evaluation questionnaires.

DETAILED DESCRIPTION:
Bone conduction hearing systems use the body's natural ability to transfer sound through bone conduction. The sound processor picks up sound and converts it into vibrations that are transferred through the skull bone to the inner ear (cochlea). Thus, for patients with conductive or mixed hearing losses, patients with lasting hearing loss following a middle ear disease or malformations (such as microtia), the vibrations are bypassing the conductive problem in the ear canal or middle ear. Bone conduction devices currently on the market are divided into three types; transcutaneous direct drive, percutaneous (skin penetrating) direct drive and transcutaneous skin drive bone conduction devices. This evaluation focus on a sound processor used for a transcutaneous system.

ELIGIBILITY:
Inclusion Criteria:

* Subjects implanted with the Bridging Bone Conductor (BBC) implant
* Subjects that have completed one year follow up in Osseofon BCI (Bone Conduction Implant) study
* Subjects available for 6 months study procedures without affecting the follow ups in the Osseofon BCI study
* Active user of the BCI SP

Exclusion Criteria:

* Inability to participate in follow-ups
* Unsuitable as judged by the principle investigator or the sub-investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2018-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Måns Eeg Olofsson, MD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- ENT departement, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Fusion Sound Processor: The group is fitted with a Fusion Sound Processor. The sound processor picks up the sound and transfer it to the implant that convert the sound to vibrations that are transmitted to the inner ear.
Period: Overall Study
Arm/Group | Fusion Sound Processor
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fusion Sound Processor
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 46.7 [22 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 10

OUTCOME MEASURES:

1. Primary Outcome: Aided Thresholds Fusion-unaided PTA
Description: Difference between Fusion-aided and unaided sound field Pure Tone Average of thresholds of frequencies 500, 1000, 2000 and 4000 Hz (PTA 4)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Fusion Sound Processor
Number analyzed (Participants) | 10
dB | 29.6 (4.4)

2. Secondary Outcome: Aided Thresholds Fusion-unaided
Description: Difference between Fusion-aided and unaided sound field Pure Tone thresholds at frequencies 250, 500, 750, 1000, 1500, 2000, 3000, 4000, 6000 and 8000 Hz
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Fusion Sound Processor
Number analyzed (Participants) | 10
dB
  250 | 10.05 (5.5)
  500 | 26.5 (7.5)
  750 | 36.5 (5.3)
  1000 | 38.0 (7.9)
  1500 | 28.5 (6.7)
  2000 | 27.5 (8.2)
  3000 | 25.0 (8.2)
  4000 | 26.5 (7.8)
  6000 | 22.5 (8.6)
  8000 | 17.5 (10.1)

3. Secondary Outcome: Aided Thresholds Fusion PTA4
Description: Difference between Fusion-aided sound field PTA4, the average for frequencies 500, 1000, 2000 and 4000 Hz (PTA 4)
Time Frame: Baseline, 1 and 6 month(s)
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Fusion Sound Processor
Number analyzed (Participants) | 10
dB
  Difference between 0-1 months | -0.290 (1.386)
  Difference between 0-6 months | -1.07 (2.93)
  Difference between 1-6 months | -0.78 (2.754)

4. Secondary Outcome: Aided Thresholds Fusion
Description: Difference between Fusion-aided sound field pure tones at frequencies 250, 500, 750, 1000, 1500, 2000, 3000, 4000, 6000 and 8000 Hz at
Time Frame: Baseline, 1 and 6 month(s)
Reporting Status: Not Posted

5. Secondary Outcome: Aided Thresholds Fusion-BCI PTA4
Description: Difference between Fusion-aided and BCI-aided sound field Pure Tone Average 4 at frequencies 500, 1000, 2000 and 4000 Hz (PTA4)
Time Frame: 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Aided Thresholds Fusion-BCI
Description: Difference between Fusion-aided and BCI-aided sound field pure tones at frequencies 250, 500, 750, 1000, 1500, 2000, 3000, 4000, 6000 and 8000 Hz
Time Frame: 6 months
Reporting Status: Not Posted

7. Secondary Outcome: Speech Intelligibility Fusion-unaided %
Description: Difference between Fusion-aided and unaided speech intelligibility scores (in % correct). Score indicates number of word repeated correctly with aided with the Fusion sound processor compared to unaided. Ranges from 0-100, a higher score indicates better performance. No scale is used.
Time Frame: 6 months
Reporting Status: Not Posted

8. Secondary Outcome: Speech Intelligibility Fusion-unaided Signal to Noise Ratio (SNR)
Description: Difference between Fusion-aided and unaided sound field speech intelligibility scores in SNR. Score indicates the signal to noise ratio where the subject can repeat 50% of the words correct. A lower score means a better outcome. No scale is used.
Time Frame: 6 months
Reporting Status: Not Posted

9. Secondary Outcome: Speech Intelligibility Fusion %
Description: Difference between Fusion-aided speech intelligibility scores (in % correct). Score indicates number of word repeated correctly with aided with the Fusion sound processor compared to unaided. Ranges from 0-100, a higher score indicates better performance. No scale is used.
Time Frame: Baseline, 1 and 6 month(s)
Reporting Status: Not Posted

10. Secondary Outcome: Speech Intelligibility Fusion SNR
Description: Difference between Fusion-aided sound field sound field speech intelligibility scores in SNR. Score indicates the signal to noise ratio where the subject can repeat 50% of the words correct. A lower score means a better outcome. No scale is used.
Time Frame: Baseline, 1 and 6 month(s)
Reporting Status: Not Posted

11. Secondary Outcome: Speech Intelligibility Fusion-BCI %
Description: Difference between Fusion-aided BCI-aided speech intelligibility scores (in % correct). Score indicates number of word repeated correctly with aided with the Fusion sound processor compared to unaided. Ranges from 0-100, a higher score indicates better performance. No scale is used
Time Frame: 6 months
Reporting Status: Not Posted

12. Secondary Outcome: Speech Intelligibility Fusion-BCI SNR
Description: Difference between Fusion-aided and BCI-aided sound field speech intelligibility scores in SNR. Score indicates the signal to noise ratio where the subject can repeat 50% of the words correct. A lower score means a better outcome. No scale is used.
Time Frame: 6 months
Reporting Status: Not Posted

13. Secondary Outcome: Magnet Strength
Description: Difference in magnet strength measured on the patient's heads in Newton
Time Frame: Baseline, 1 and 6 month(s)
Reporting Status: Not Posted

14. Secondary Outcome: IPS (Inflammation, Pain, Skin Height/Numbness) Evaluation
Description: Combined score of IInflammation, Pain and Skin height/numbness scale evaluating the skin area under the sound processor. I scale ranging from 0-4, Pain scale ranging from 0-2, Skin height/numbness ranging from 0-2. Total score 0-8 (0 no adverse skin condition, 8 maximum adverse skin reactions on all subscales). Lower score means better performance
Time Frame: Baseline, 1 and 6 month(s)
Reporting Status: Not Posted

15. Secondary Outcome: Subjective Evaluation
Description: User satisfaction and usability as measured with questionniare "Usage of sound processor" consisting of rating scales on satisfaction of the sound processor. The scale used is a scale with descriptive values.
Time Frame: Baseline, 1 and 6 month(s)
Reporting Status: Not Posted

16. Secondary Outcome: Subjective Evaluation SSQ
Description: Subjective performance as measured by Speech, Spatial and Qualities of hearing (SSQ) a scale from 0-10 where 0 represents "Not at all" and 10 represents "Perfect". A higher score means better performance.
Time Frame: Baseline, 1 and 6 month(s)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Fusion Sound Processor
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 7/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fusion Sound Processor (N=10)
Implant site pain (General disorders) | 1 (1)
Implat site paraesthesia (General disorders) | 1 (1)
Medical device site irritation (General disorders) | 1 (1)
Pyrexia (General disorders) | 1
Seasonal allergy (Immune system disorders) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-04): https://cdn.clinicaltrials.gov/large-docs/87/NCT03374787/Prot_SAP_000.pdf